CLINICAL TRIAL: NCT02849782
Title: Short and Long Term Fampridine Treatment in Persons With Multiple Sclerosis: Cognitive and Motor Performances
Brief Title: Short and Long Term Multiple Outcomes in Persons With Multiple Sclerosis Treated by Fampridine.
Acronym: FAMPISEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: API/2014/49
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
Keywords: Gait analysis; Fampridine; Fatigue; Daily activity; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fampridine responder (Experimental): Persons who have been diagnosed as Multiple Sclerosis according to Mc Donald Criteria : person with Multiple Sclerosis (PwMS).
  Fampridine was prescribed according to the guidelines issued by the French National Security Agency of Medicines and Health Products (ANSM) at the dose of 10 mg twice a day. According to official ANSM guidelines, the prescription is initially limited to 2 weeks of therapy, at which point a new assessment is performed by the medical practitioner to evaluate the clinical benefits. Fampridine responder is a PwMS with an improvement in the judgment of the practitioner.
  Interventions: Drug: Fampridine
- Fampridine non responder (Active Comparator): Persons who have been diagnosed as Multiple Sclerosis according to Mc Donald Criteria : person with Multiple Sclerosis (PwMS).
  Fampridine was prescribed according to the guidelines issued by the French National Security Agency of Medicines and Health Products (ANSM) at the dose of 10 mg twice a day. According to official ANSM guidelines, the prescription is initially limited to 2 weeks of therapy, at which point a new assessment is performed by the medical practitioner to evaluate the clinical benefits. Fampridine non responder is a PwMS without any improvement in the judgment of the practitioner.
  Interventions: Drug: Fampridine

INTERVENTIONS:
Drug: Fampridine — Oral intake of 10 mg twice daily
  Other Names: Fampyra; code CIS : 62483787

SUMMARY:
This prospective monocentric open label trial was realized in the Laboratory of Clinical Functional Exploration of Movement at the University Hospital of Besancon. Cognitive evaluations: 7 days before fampridine treatment initiation (Pre 1), on the day of fampridine treatment initiation (Pre 2), 14 and 21 days after fampridine treatment initiation, respectively Post 1 and Post 2. Gait evaluations were assessed at Pre 1, Pre 2 and Post 1.

Fampridine was prescribed according to guidelines issued by the French Health Products Safety Agency at the dose of 10 mg twice daily. Fampridine is indicated for the improvement of walking in MS patients with a walking disability (EDSS 4-6.5). A walking test is recommended to evaluate improvement after 2 weeks of treatment. According to the practitioner evaluation between Pre 2 and Post 1 (i.e. before and after fampridine treatment), patients were classified into 2 groups: responders whose clinical status was improved and non-responders whose clinical status was not improved.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic neurological disorder affecting young and middle-aged adults with a female to male ratio of more than 3:1. The cause of MS is unknown although it involves genetic susceptibility and environmental exposure. Since there is no known cure for MS, the main goals of treatment is to delay progression of the disease and to improve health-related quality of life (HRQoL) by masking patients' symptoms. Among several symptoms of MS (e.g., motor and cognitive impairments, optic neuritis, fatigue, pain, urinary dysfunction), gait impairment, defined as an activity limitation by the International Classification of Functioning Disability and Health, is one of the most common and disabling dysfunction in Persons with Multiple Sclerosis PwMS. Studies have reported that approximately 75 % of individuals with MS experience clinically significant walking disturbances. Likewise, fatigue, impairment of information-processing speed (IPS), attention, working memory and executive functions can occur in MS and can worsen during the evolution of the disease.

Studies have shown that MS symptomatic treatment by fampridine (4-aminopyridine) is associated with improvements in walking and muscle strength and possibly with cognition, vision, fatigue and spasticity. Indeed, fampridine is a potassium channel blocker which reduces the leakage of ionic current through these channels, prolonging repolarization and thus, enhancing action-potential formation in demyelinated axons. Presumably, by enhancing action-potential formation, more impulses might be conducted in the central nervous system (CNS) and neurological functions could be ameliorated. In recent phase III studies, Goodman et al. investigated the fampridine effect on the walk of individuals with MS during a timed 25-foot walk test (T25FW). Improvement in walking velocity (≈25 % from baseline) was found for 35-43 % of the individuals in the interventional group.

However, improvement in neuronal conduction induced by fampridine might not be limited to short distances of gait or even to motor functions and might also improve long distance ambulation or cognitive functions.

Different assessments have been used for measuring gait impairments in multiple sclerosis, including the Timed 25-Foot Walk (T25FW), Six-Minute Walk Test (6MWT), spatio-temporal gait parameters measured with an instrumented walkway or the Timed Up and Go test (TUG). These different assessments can be performed at different conditions: simple task, fast speed or dual task. In this last case, the gait is associated with a cognitive or another motor task. For cognitive assessments, Symbol Digit Modalities Test (SDMT) and verbal fluencies have been used in previous studies.

The aimed of the study was to evaluate the impact of fampridine in gait evaluating by long distance tests and to evaluate the impact of fampridine in fatigue and cognition.

Assessments of patients were performed 7 days before fampridine treatment initiation (Pre 1), on the day of fampridine treatment initiation (Pre 2), 14 and 21 days after fampridine treatment initiation, respectively Post 1 and Post 2. Gait evaluations were assessed at Pre 1, Pre 2 and Post 1. The first two assessments were intended to evaluate the variability of measurement without any treatment. A measurement of activity was performed by accelerometer during the period covering the first two assessments. The third assessment was intend to measure clinical improvements. The fourth seeks to show a potentially delayed action of fampridine on cognition.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnostic regarding the modified McDonald criteria
* EDSS status between 4.0 and 6.5
* patients able to walk during 6 minutes

Exclusion Criteria:

* increasing MS symptoms during the previous 60 days
* history of epilepsy or epileptic seizure
* immunotherapy change in the previous 60 days
* beginning anti-spastic treatment in the previous 30 days
* beginning treatment that is able to decrease fatigue symptoms in the previous 30 days
* modification of the rehabilitation program during the study
* renal insufficiency (creatinine clearance <80ml.min-1 given by the Cockroft-Gault formula)
* concomitant treatment by organic cation transporter 2 inhibitor
* hypersensitivity to fampridine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | Timed 21 days
  The 6MWT assessed the submaximal level of functional capacity. It was realized according to the recommendation of the American Thoracic Society. 6MWT instructions were read prior to each walk. Participants used his/her typical assistive device and walked around a circuit with 24-meters longer. If necessary, they were allowed to have a rest period and encouragement phrases were used each 30 seconds.

SECONDARY OUTCOMES:
Verbal fluencies | Day 1
  Both semantic and phonological verbal fluencies were assessed in a quiet room. Semantic fluency was measured by asking patients to provide as many animal names as possible in 120 s. Different kinds of one sort of animal were accepted (e.g. kinds of birds or fish). Phonological fluency was measured by asking patients to provide as many words as possible beginning with the letter 'P' in 120 s. They were informed that proper nouns and words with the same stem would not be counted (e.g. pen, pencil). Patients were instructed to avoid repetitions.
Verbal fluencies | 7 days
  Both semantic and phonological verbal fluencies were assessed in a quiet room. Semantic fluency was measured by asking patients to provide as many animal names as possible in 120 s. Different kinds of one sort of animal were accepted (e.g. kinds of birds or fish). Phonological fluency was measured by asking patients to provide as many words as possible beginning with the letter 'P' in 120 s. They were informed that proper nouns and words with the same stem would not be counted (e.g. pen, pencil). Patients were instructed to avoid repetitions.
Verbal fluencies | 21 days
  Both semantic and phonological verbal fluencies were assessed in a quiet room. Semantic fluency was measured by asking patients to provide as many animal names as possible in 120 s. Different kinds of one sort of animal were accepted (e.g. kinds of birds or fish). Phonological fluency was measured by asking patients to provide as many words as possible beginning with the letter 'P' in 120 s. They were informed that proper nouns and words with the same stem would not be counted (e.g. pen, pencil). Patients were instructed to avoid repetitions.
Verbal fluencies | 28 days
  Both semantic and phonological verbal fluencies were assessed in a quiet room. Semantic fluency was measured by asking patients to provide as many animal names as possible in 120 s. Different kinds of one sort of animal were accepted (e.g. kinds of birds or fish). Phonological fluency was measured by asking patients to provide as many words as possible beginning with the letter 'P' in 120 s. They were informed that proper nouns and words with the same stem would not be counted (e.g. pen, pencil). Patients were instructed to avoid repetitions.
Verbal fluencies | up to one year
  Both semantic and phonological verbal fluencies were assessed in a quiet room. Semantic fluency was measured by asking patients to provide as many animal names as possible in 120 s. Different kinds of one sort of animal were accepted (e.g. kinds of birds or fish). Phonological fluency was measured by asking patients to provide as many words as possible beginning with the letter 'P' in 120 s. They were informed that proper nouns and words with the same stem would not be counted (e.g. pen, pencil). Patients were instructed to avoid repetitions.
Symbol Digit Modalities Test | Day 1
  The SDMT has a key at the top of the page with numbers and symbols; participants are required to refer to the key to correctly decode several lines of symbols. After completing sample items correctly, participants are timed for 90 s and the total number correct is their raw score. Only correct answers were account to the final score.
Symbol Digit Modalities Test | 7 days
  The SDMT has a key at the top of the page with numbers and symbols; participants are required to refer to the key to correctly decode several lines of symbols. After completing sample items correctly, participants are timed for 90 s and the total number correct is their raw score. Only correct answers were account to the final score.
Symbol Digit Modalities Test | 21 days
  The SDMT has a key at the top of the page with numbers and symbols; participants are required to refer to the key to correctly decode several lines of symbols. After completing sample items correctly, participants are timed for 90 s and the total number correct is their raw score. Only correct answers were account to the final score.
Symbol Digit Modalities Test | 28 days
  The SDMT has a key at the top of the page with numbers and symbols; participants are required to refer to the key to correctly decode several lines of symbols. After completing sample items correctly, participants are timed for 90 s and the total number correct is their raw score. Only correct answers were account to the final score.
Symbol Digit Modalities Test | up to one year
  The SDMT has a key at the top of the page with numbers and symbols; participants are required to refer to the key to correctly decode several lines of symbols. After completing sample items correctly, participants are timed for 90 s and the total number correct is their raw score. Only correct answers were account to the final score.
Modified Fatigue Impact Scale (mFIS) | day 1
  The FIS is a 40-item Standardized questionnaire validated for MS. For our study, we used the validated French version of the FIS in MS, called "EMIF-SEP". The EMIF-SEP is composed of 40 items organized into four dimensions (cognitive, physical, social role and psychological dimensions) with each items rated on a four point scale (4=it's always true, 3=it's sometimes true, 2=it's sometimes false, 1=it's always false) and the total fatigue scores are standardized from 0 (meaning no fatigue) to 100 (meaning high degree of fatigue). The forty items are divided into the four dimensions: cognitive (10 items), physical (14 items), social role (13 items) and psychological (4 items). Each dimension score was also standardized as a percentage like total score.
Modified Fatigue Impact Scale (mFIS) | 7 days
  The FIS is a 40-item Standardized questionnaire validated for MS. For our study, we used the validated French version of the FIS in MS, called "EMIF-SEP". The EMIF-SEP is composed of 40 items organized into four dimensions (cognitive, physical, social role and psychological dimensions) with each items rated on a four point scale (4=it's always true, 3=it's sometimes true, 2=it's sometimes false, 1=it's always false) and the total fatigue scores are standardized from 0 (meaning no fatigue) to 100 (meaning high degree of fatigue). The forty items are divided into the four dimensions: cognitive (10 items), physical (14 items), social role (13 items) and psychological (4 items). Each dimension score was also standardized as a percentage like total score.
Modified Fatigue Impact Scale (mFIS) | 21 days
  The FIS is a 40-item Standardized questionnaire validated for MS. For our study, we used the validated French version of the FIS in MS, called "EMIF-SEP". The EMIF-SEP is composed of 40 items organized into four dimensions (cognitive, physical, social role and psychological dimensions) with each items rated on a four point scale (4=it's always true, 3=it's sometimes true, 2=it's sometimes false, 1=it's always false) and the total fatigue scores are standardized from 0 (meaning no fatigue) to 100 (meaning high degree of fatigue). The forty items are divided into the four dimensions: cognitive (10 items), physical (14 items), social role (13 items) and psychological (4 items). Each dimension score was also standardized as a percentage like total score.
Modified Fatigue Impact Scale (mFIS) | 28 days
  The FIS is a 40-item Standardized questionnaire validated for MS. For our study, we used the validated French version of the FIS in MS, called "EMIF-SEP". The EMIF-SEP is composed of 40 items organized into four dimensions (cognitive, physical, social role and psychological dimensions) with each items rated on a four point scale (4=it's always true, 3=it's sometimes true, 2=it's sometimes false, 1=it's always false) and the total fatigue scores are standardized from 0 (meaning no fatigue) to 100 (meaning high degree of fatigue). The forty items are divided into the four dimensions: cognitive (10 items), physical (14 items), social role (13 items) and psychological (4 items). Each dimension score was also standardized as a percentage like total score.
Modified Fatigue Impact Scale (mFIS) | up to one year
  The FIS is a 40-item Standardized questionnaire validated for MS. For our study, we used the validated French version of the FIS in MS, called "EMIF-SEP". The EMIF-SEP is composed of 40 items organized into four dimensions (cognitive, physical, social role and psychological dimensions) with each items rated on a four point scale (4=it's always true, 3=it's sometimes true, 2=it's sometimes false, 1=it's always false) and the total fatigue scores are standardized from 0 (meaning no fatigue) to 100 (meaning high degree of fatigue). The forty items are divided into the four dimensions: cognitive (10 items), physical (14 items), social role (13 items) and psychological (4 items). Each dimension score was also standardized as a percentage like total score.
Fatigue Severity Scale (FSS) | day 1
  The FSS is a method of evaluating fatigue in PwMS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus. The FSS is designed to differentiate fatigue from clinical depression because both share some of the same symptoms. The FSS questionnaire is composed of 9 statements related to patients' subjective perception of fatigue and its consequences on everyday activities. Patients are asked to rate their level of agreement (toward 7) or disagreement (toward 0) with the 9 statements.
Fatigue Severity Scale (FSS) | 7 days
  The FSS is a method of evaluating fatigue in PwMS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus. The FSS is designed to differentiate fatigue from clinical depression because both share some of the same symptoms. The FSS questionnaire is composed of 9 statements related to patients' subjective perception of fatigue and its consequences on everyday activities. Patients are asked to rate their level of agreement (toward 7) or disagreement (toward 0) with the 9 statements.
Fatigue Severity Scale (FSS) | 21 days
  The FSS is a method of evaluating fatigue in PwMS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus. The FSS is designed to differentiate fatigue from clinical depression because both share some of the same symptoms. The FSS questionnaire is composed of 9 statements related to patients' subjective perception of fatigue and its consequences on everyday activities. Patients are asked to rate their level of agreement (toward 7) or disagreement (toward 0) with the 9 statements.
Fatigue Severity Scale (FSS) | 28 days
  The FSS is a method of evaluating fatigue in PwMS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus. The FSS is designed to differentiate fatigue from clinical depression because both share some of the same symptoms. The FSS questionnaire is composed of 9 statements related to patients' subjective perception of fatigue and its consequences on everyday activities. Patients are asked to rate their level of agreement (toward 7) or disagreement (toward 0) with the 9 statements.
Fatigue Severity Scale (FSS) | up to one year
  The FSS is a method of evaluating fatigue in PwMS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus. The FSS is designed to differentiate fatigue from clinical depression because both share some of the same symptoms. The FSS questionnaire is composed of 9 statements related to patients' subjective perception of fatigue and its consequences on everyday activities. Patients are asked to rate their level of agreement (toward 7) or disagreement (toward 0) with the 9 statements.
Multiple Sclerosis Walking Scale 12 (MSWS12) | day 1
  The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
Multiple Sclerosis Walking Scale 12 (MSWS12) | 7 days
  The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
Multiple Sclerosis Walking Scale 12 (MSWS12) | 21 days
  The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
Multiple Sclerosis Walking Scale 12 (MSWS12) | 28 days
  The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
Multiple Sclerosis Walking Scale 12 (MSWS12) | up to one year
  The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
"PERception de la Sclérose En Plaques et de ses Poussées" (PERSEPP) | day 1
  The PERSEPP scale was used to evaluate the HRQoL of patients with MS (Baroin et al. 2013). This scale takes into account several aspects of HRQoL distributed across 66 items (described below) and includes relapse phases. Each item contains 6 response types according to a Likert scale where "0" was "strongly disagree" and "5" was "strongly agree". The PERSEPP scale has been validated in the French language
"PERception de la Sclérose En Plaques et de ses Poussées" (PERSEPP) | day 7
  The PERSEPP scale was used to evaluate the HRQoL of patients with MS (Baroin et al. 2013). This scale takes into account several aspects of HRQoL distributed across 66 items (described below) and includes relapse phases. Each item contains 6 response types according to a Likert scale where "0" was "strongly disagree" and "5" was "strongly agree". The PERSEPP scale has been validated in the French language
"PERception de la Sclérose En Plaques et de ses Poussées" (PERSEPP) | day 21
  The PERSEPP scale was used to evaluate the HRQoL of patients with MS (Baroin et al. 2013). This scale takes into account several aspects of HRQoL distributed across 66 items (described below) and includes relapse phases. Each item contains 6 response types according to a Likert scale where "0" was "strongly disagree" and "5" was "strongly agree". The PERSEPP scale has been validated in the French language
"PERception de la Sclérose En Plaques et de ses Poussées" (PERSEPP) | day 28
  The PERSEPP scale was used to evaluate the HRQoL of patients with MS (Baroin et al. 2013). This scale takes into account several aspects of HRQoL distributed across 66 items (described below) and includes relapse phases. Each item contains 6 response types according to a Likert scale where "0" was "strongly disagree" and "5" was "strongly agree". The PERSEPP scale has been validated in the French language
"PERception de la Sclérose En Plaques et de ses Poussées" (PERSEPP) | up to one year
  The PERSEPP scale was used to evaluate the HRQoL of patients with MS (Baroin et al. 2013). This scale takes into account several aspects of HRQoL distributed across 66 items (described below) and includes relapse phases. Each item contains 6 response types according to a Likert scale where "0" was "strongly disagree" and "5" was "strongly agree". The PERSEPP scale has been validated in the French language
Physical activity in real life condition | During 7 days (day 1 to day 7)
  The physical activity in real-life condition was measured with an ActiGraph, model wGT3X (Actigraph corp, USA), consistent with previous research on validating accelerometer output in PwMS. The accelerometer was sampled at 30 Hz and values were expressed as number of counts per minute. Participants were instructed to wear the accelerometer on an elastic belt around the waist (i.e. near to the center of displacement of body mass) located above the hip at the non-dominant side ; to wear it for a 7-day period (including a weekend); and to wear it for the whole day from getting out of bed in the morning until getting into bed in the evening. These instructions were summarized in a memo and given to participants.
Physical activity in real life condition | During 7 days (day 21 to day 28)
  The physical activity in real-life condition was measured with an ActiGraph, model wGT3X (Actigraph corp, USA), consistent with previous research on validating accelerometer output in PwMS. The accelerometer was sampled at 30 Hz and values were expressed as number of counts per minute. Participants were instructed to wear the accelerometer on an elastic belt around the waist (i.e. near to the center of displacement of body mass) located above the hip at the non-dominant side ; to wear it for a 7-day period (including a weekend); and to wear it for the whole day from getting out of bed in the morning until getting into bed in the evening. These instructions were summarized in a memo and given to participants.
Timed 25 Walk Test (T25WT) | Day 1
  According with the recommendation of Cutter et al., participants were asked to walk on a 25 feet (7.62 m) distance. After appropriate instructions and familiarization, participants were asked to perform three gait tasks: walking at their self-selected comfortable speed .
Timed 25 Walk Test (T25WT) | 7 days
  According with the recommendation of Cutter et al., participants were asked to walk on a 25 feet (7.62 m) distance. After appropriate instructions and familiarization, participants were asked to perform three gait tasks: walking at their self-selected comfortable speed .
Timed 25 Walk Test (T25WT) | 21 days
  According with the recommendation of Cutter et al., participants were asked to walk on a 25 feet (7.62 m) distance. After appropriate instructions and familiarization, participants were asked to perform three gait tasks: walking at their self-selected comfortable speed .
Timed 25 Walk Test (T25WT) | 28 days
  According with the recommendation of Cutter et al., participants were asked to walk on a 25 feet (7.62 m) distance. After appropriate instructions and familiarization, participants were asked to perform three gait tasks: walking at their self-selected comfortable speed .
Timed 25 Walk Test (T25WT) | up to one year
  According with the recommendation of Cutter et al., participants were asked to walk on a 25 feet (7.62 m) distance. After appropriate instructions and familiarization, participants were asked to perform three gait tasks: walking at their self-selected comfortable speed .
Timed Up and Go test (TUG) | Day 1
  The TUG is a clinical test to assess the level of gait and balance. For its realization, a 47-cm-high chair with arm- and backrest was used. The 3-meters distance was marked with a tape on the floor and a cone marked the turning point. Participants were instructed to get up from the chair, walk 3 meters, turn around the cone and come back to sit on the chair. Participants were encouraged to walk as quickly as possible with safety consistency. After a familiarization trial, the TUG was performed twice. A third trial was applied if a difference of 10% was found between the two first trials. The mean value computed from the two closest trials was taken into account.
Timed Up and Go test (TUG) | 7 days
  The TUG is a clinical test to assess the level of gait and balance. For its realization, a 47-cm-high chair with arm- and backrest was used. The 3-meters distance was marked with a tape on the floor and a cone marked the turning point. Participants were instructed to get up from the chair, walk 3 meters, turn around the cone and come back to sit on the chair. Participants were encouraged to walk as quickly as possible with safety consistency. After a familiarization trial, the TUG was performed twice. A third trial was applied if a difference of 10% was found between the two first trials. The mean value computed from the two closest trials was taken into account.
Timed Up and Go test (TUG) | 21
  The TUG is a clinical test to assess the level of gait and balance. For its realization, a 47-cm-high chair with arm- and backrest was used. The 3-meters distance was marked with a tape on the floor and a cone marked the turning point. Participants were instructed to get up from the chair, walk 3 meters, turn around the cone and come back to sit on the chair. Participants were encouraged to walk as quickly as possible with safety consistency. After a familiarization trial, the TUG was performed twice. A third trial was applied if a difference of 10% was found between the two first trials. The mean value computed from the two closest trials was taken into account.
Timed Up and Go test (TUG) | 28 days
  The TUG is a clinical test to assess the level of gait and balance. For its realization, a 47-cm-high chair with arm- and backrest was used. The 3-meters distance was marked with a tape on the floor and a cone marked the turning point. Participants were instructed to get up from the chair, walk 3 meters, turn around the cone and come back to sit on the chair. Participants were encouraged to walk as quickly as possible with safety consistency. After a familiarization trial, the TUG was performed twice. A third trial was applied if a difference of 10% was found between the two first trials. The mean value computed from the two closest trials was taken into account.
Timed Up and Go test (TUG) | up to one year
  The TUG is a clinical test to assess the level of gait and balance. For its realization, a 47-cm-high chair with arm- and backrest was used. The 3-meters distance was marked with a tape on the floor and a cone marked the turning point. Participants were instructed to get up from the chair, walk 3 meters, turn around the cone and come back to sit on the chair. Participants were encouraged to walk as quickly as possible with safety consistency. After a familiarization trial, the TUG was performed twice. A third trial was applied if a difference of 10% was found between the two first trials. The mean value computed from the two closest trials was taken into account.
6 Minute Walk Test (6MWT) | day 1
  The 6MWT assessed the submaximal level of functional capacity. It was realized according to the recommendation of the American Thoracic Society. 6MWT instructions were read prior to each walk. Participants used his/her typical assistive device and walked around a circuit with 24-meters longer. If necessary, they were allowed to have a rest period and encouragement phrases were used each 30 seconds.
6 Minute Walk Test (6MWT) | day 7
  The 6MWT assessed the submaximal level of functional capacity. It was realized according to the recommendation of the American Thoracic Society. 6MWT instructions were read prior to each walk. Participants used his/her typical assistive device and walked around a circuit with 24-meters longer. If necessary, they were allowed to have a rest period and encouragement phrases were used each 30 seconds.
6 Minute Walk Test (6MWT) | day 28
  The 6MWT assessed the submaximal level of functional capacity. It was realized according to the recommendation of the American Thoracic Society. 6MWT instructions were read prior to each walk. Participants used his/her typical assistive device and walked around a circuit with 24-meters longer. If necessary, they were allowed to have a rest period and encouragement phrases were used each 30 seconds.
6 Minute Walk Test (6MWT) | up to one year
  The 6MWT assessed the submaximal level of functional capacity. It was realized according to the recommendation of the American Thoracic Society. 6MWT instructions were read prior to each walk. Participants used his/her typical assistive device and walked around a circuit with 24-meters longer. If necessary, they were allowed to have a rest period and encouragement phrases were used each 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Jean Minjoz, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allart E, Benoit A, Blanchard-Dauphin A, Tiffreau V, Thevenon A, Zephir H, Outteryck O, Lacour A, Vermersch P. Sustained-released fampridine in multiple sclerosis: effects on gait parameters, arm function, fatigue, and quality of life. J Neurol. 2015 Aug;262(8):1936-45. doi: 10.1007/s00415-015-7797-1. Epub 2015 Jun 5. PMID 26041616
- [Result] Almarwani M, Perera S, VanSwearingen JM, Sparto PJ, Brach JS. The test-retest reliability and minimal detectable change of spatial and temporal gait variability during usual over-ground walking for younger and older adults. Gait Posture. 2016 Feb;44:94-9. doi: 10.1016/j.gaitpost.2015.11.014. Epub 2015 Nov 30. PMID 27004639
- [Result] Baert I, Freeman J, Smedal T, Dalgas U, Romberg A, Kalron A, Conyers H, Elorriaga I, Gebara B, Gumse J, Heric A, Jensen E, Jones K, Knuts K, Maertens de Noordhout B, Martic A, Normann B, Eijnde BO, Rasova K, Santoyo Medina C, Truyens V, Wens I, Feys P. Responsiveness and clinically meaningful improvement, according to disability level, of five walking measures after rehabilitation in multiple sclerosis: a European multicenter study. Neurorehabil Neural Repair. 2014 Sep;28(7):621-31. doi: 10.1177/1545968314521010. Epub 2014 Feb 6. PMID 24503204
- [Result] Baroin A, Chopard G, Siliman G, Michoudet C, Vivot A, Vidal C, Mokadym H, Lavier A, Berger E, Rumbach L, Rude N. Validation of a new quality of life scale related to multiple sclerosis and relapses. Qual Life Res. 2013 Oct;22(8):1943-54. doi: 10.1007/s11136-012-0334-0. Epub 2012 Dec 18. PMID 23247892
- [Result] Bland JM, Altman DG. Measurement error. BMJ. 1996 Jun 29;312(7047):1654. doi: 10.1136/bmj.312.7047.1654. No abstract available. PMID 8664723
- [Result] Brochet B, Deloire MS, Bonnet M, Salort-Campana E, Ouallet JC, Petry KG, Dousset V. Should SDMT substitute for PASAT in MSFC? A 5-year longitudinal study. Mult Scler. 2008 Nov;14(9):1242-9. doi: 10.1177/1352458508094398. Epub 2008 Jul 24. PMID 18653737
- [Result] Confavreux C, Vukusic S. The clinical epidemiology of multiple sclerosis. Neuroimaging Clin N Am. 2008 Nov;18(4):589-622, ix-x. doi: 10.1016/j.nic.2008.09.002. PMID 19068404
- [Result] Debouverie M, Pittion-Vouyovitch S, Louis S, Guillemin F. Validity of a French version of the fatigue impact scale in multiple sclerosis. Mult Scler. 2007 Sep;13(8):1026-32. doi: 10.1177/1352458507077942. PMID 17895294
- [Result] de Vet HC, Terwee CB, Knol DL, Bouter LM. When to use agreement versus reliability measures. J Clin Epidemiol. 2006 Oct;59(10):1033-9. doi: 10.1016/j.jclinepi.2005.10.015. Epub 2006 Aug 10. PMID 16980142
- [Result] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Result] Givon U, Zeilig G, Achiron A. Gait analysis in multiple sclerosis: characterization of temporal-spatial parameters using GAITRite functional ambulation system. Gait Posture. 2009 Jan;29(1):138-42. doi: 10.1016/j.gaitpost.2008.07.011. Epub 2008 Oct 31. PMID 18951800
- [Result] Goldman MD, Marrie RA, Cohen JA. Evaluation of the six-minute walk in multiple sclerosis subjects and healthy controls. Mult Scler. 2008 Apr;14(3):383-90. doi: 10.1177/1352458507082607. Epub 2007 Oct 17. PMID 17942508
- [Result] Goodkin DE. EDSS reliability. Neurology. 1991 Feb;41(2 ( Pt 1)):332. doi: 10.1212/wnl.41.2_part_1.332. No abstract available. PMID 1992392
- [Result] Goodman AD, Bethoux F, Brown TR, Schapiro RT, Cohen R, Marinucci LN, Henney HR 3rd, Blight AR; MS-F203, MS-F204, and Extension Study Investigators. Long-term safety and efficacy of dalfampridine for walking impairment in patients with multiple sclerosis: Results of open-label extensions of two Phase 3 clinical trials. Mult Scler. 2015 Sep;21(10):1322-31. doi: 10.1177/1352458514563591. Epub 2015 Jan 12. PMID 25583832
- [Result] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- [Result] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Result] Hobart J, Blight AR, Goodman A, Lynn F, Putzki N. Timed 25-foot walk: direct evidence that improving 20% or greater is clinically meaningful in MS. Neurology. 2013 Apr 16;80(16):1509-17. doi: 10.1212/WNL.0b013e31828cf7f3. Epub 2013 Mar 27. PMID 23535489
- [Result] Kalron A, Dvir Z, Achiron A. Walking while talking--difficulties incurred during the initial stages of multiple sclerosis disease process. Gait Posture. 2010 Jul;32(3):332-5. doi: 10.1016/j.gaitpost.2010.06.002. Epub 2010 Jul 1. PMID 20594850
- [Result] Kalron A. Gait variability across the disability spectrum in people with multiple sclerosis. J Neurol Sci. 2016 Feb 15;361:1-6. doi: 10.1016/j.jns.2015.12.012. Epub 2015 Dec 10. PMID 26810506
- [Result] Learmonth YC, Dlugonski D, Pilutti LA, Sandroff BM, Klaren R, Motl RW. Psychometric properties of the Fatigue Severity Scale and the Modified Fatigue Impact Scale. J Neurol Sci. 2013 Aug 15;331(1-2):102-7. doi: 10.1016/j.jns.2013.05.023. Epub 2013 Jun 20. PMID 23791482
- [Result] Learmonth YC, Paul L, McFadyen AK, Mattison P, Miller L. Reliability and clinical significance of mobility and balance assessments in multiple sclerosis. Int J Rehabil Res. 2012 Mar;35(1):69-74. doi: 10.1097/MRR.0b013e328350b65f. PMID 22315143
- [Result] Moon Y, Wajda DA, Motl RW, Sosnoff JJ. Stride-Time Variability and Fall Risk in Persons with Multiple Sclerosis. Mult Scler Int. 2015;2015:964790. doi: 10.1155/2015/964790. Epub 2015 Dec 30. PMID 26843986
- [Result] Motl RW, Dlugonski D, Suh Y, Weikert M, Fernhall B, Goldman M. Accelerometry and its association with objective markers of walking limitations in ambulatory adults with multiple sclerosis. Arch Phys Med Rehabil. 2010 Dec;91(12):1942-7. doi: 10.1016/j.apmr.2010.08.011. PMID 21112438
- [Result] Motl RW, Sosnoff JJ, Dlugonski D, Pilutti LA, Klaren R, Sandroff BM. Walking and cognition, but not symptoms, correlate with dual task cost of walking in multiple sclerosis. Gait Posture. 2014 Mar;39(3):870-4. doi: 10.1016/j.gaitpost.2013.11.023. Epub 2013 Dec 14. PMID 24378281
- [Result] Pilutti LA, Dlugonski D, Sandroff BM, Suh Y, Pula JH, Sosnoff JJ, Motl RW. Gait and six-minute walk performance in persons with multiple sclerosis. J Neurol Sci. 2013 Nov 15;334(1-2):72-6. doi: 10.1016/j.jns.2013.07.2511. Epub 2013 Jul 30. PMID 23962697
- [Result] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Result] Sandroff BM, Pilutti LA, Motl RW. Does the six-minute walk test measure walking performance or physical fitness in persons with multiple sclerosis? NeuroRehabilitation. 2015;37(1):149-55. doi: 10.3233/NRE-151247. PMID 26409700
- [Result] van Uden CJ, Besser MP. Test-retest reliability of temporal and spatial gait characteristics measured with an instrumented walkway system (GAITRite). BMC Musculoskelet Disord. 2004 May 17;5:13. doi: 10.1186/1471-2474-5-13. PMID 15147583
- [Result] Vlaar AM, Wade DT. Verbal fluency assessment of patients with multiple sclerosis: test-retest and inter-observer reliability. Clin Rehabil. 2003 Nov;17(7):756-64. doi: 10.1191/0269215503cr674oa. PMID 14606742
- [Result] Wajda DA, Motl RW, Sosnoff JJ. Dual task cost of walking is related to fall risk in persons with multiple sclerosis. J Neurol Sci. 2013 Dec 15;335(1-2):160-3. doi: 10.1016/j.jns.2013.09.021. Epub 2013 Sep 20. PMID 24090757
- [Derived] Magnin E, Sagawa Y, Moulin T, Decavel P. What Are the Minimal Detectable Changes in SDMT and Verbal Fluency Tests for Assessing Changes in Cognitive Performance in Persons with Multiple Sclerosis and Non-Multiple Sclerosis Controls? Eur Neurol. 2020;83(3):263-270. doi: 10.1159/000508607. Epub 2020 Jul 7. PMID 32634812